CLINICAL TRIAL: NCT04489134
Title: P-glypoprotein Inhibition Effect on the Pharmacokinetics of Two Tacrolimus Formulations: Prolonged and Extended-release
Acronym: DIPLOID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 35RC19_8877_DIPLOID
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This is a pharmacokinetic, monocentric, prospective, randomized, crossover study with blind assessment (biologists performing tacrolimus dosages will be blind to the treatment received).
Who Masked: Outcomes Assessor
Masking Description: the biologists performing the tacrolimus assays will be blind to the treatment received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A D B C (Experimental): Period n°01: Administration of a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°02:Administration of a single 120 mg dose of immediate release verapamil (Isoptine®) and a 2 mg dose of LCP-tacro (Envarsus®) Period n°03:Administration of a 2 mg dose of LCP-tacro (Envarsus®) Period n°04:Administration of a single 120 mg dose of immediate-release verapamil (Isoptine®) and a 3 mg dose of prolonged-release tacrolimus (Advagraf®)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treament C; Drug: Treatment D; Biological: Pharmacocinetik; Genetic: Genetic; Other: Selection visit:
- B A C D (Experimental): Period n°01: Administration of a 2 mg dose of LCP-tacro (Envarsus®) Period n°02:Administration of a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°03:Administration of a single 120 mg dose of immediate-release verapamil (Isoptine®) and a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°04:Administration of a single 120 mg dose of immediate release verapamil (Isoptine®) and a 2 mg dose of LCP-tacro (Envarsus®)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treament C; Drug: Treatment D; Biological: Pharmacocinetik; Genetic: Genetic; Other: Selection visit:
- C B D A (Experimental): Period n°01: Administration of a single 120 mg dose of immediate-release verapamil (Isoptine®) and a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°02:Administration of a 2 mg dose of LCP-tacro (Envarsus®) Period n°03:Administration of a single 120 mg dose of immediate release verapamil (Isoptine®) and a 2 mg dose of LCP-tacro (Envarsus®) Period n°04:Administration of a 3 mg dose of prolonged-release tacrolimus (Advagraf®)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treament C; Drug: Treatment D; Biological: Pharmacocinetik; Genetic: Genetic; Other: Selection visit:
- D C A B (Experimental): Period n°01:Administration of a single 120 mg dose of immediate release verapamil (Isoptine®) and a 2 mg dose of LCP-tacro (Envarsus®) Period n°02:Administration of a single 120 mg dose of immediate-release verapamil (Isoptine®) and a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°03:Administration of a 3 mg dose of prolonged-release tacrolimus (Advagraf®) Period n°04:Administration of a 2 mg dose of LCP-tacro (Envarsus®)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treament C; Drug: Treatment D; Biological: Pharmacocinetik; Genetic: Genetic; Other: Selection visit:

INTERVENTIONS:
Drug: Treatment A — Administration of a 3 mg dose of prolonged-release tacrolimus (Advagraf®)
Drug: Treatment B — Administration of a 2 mg dose of LCP-tacro (Envarsus®)
Drug: Treament C — Administration of a single 120 mg dose of immediate-release verapamil (Isoptine®) and a 3 mg dose of prolonged-release tacrolimus (Advagraf®)
Drug: Treatment D — Administration of a single 120 mg dose of immediate release verapamil (Isoptine®) and a 2 mg dose of LCP-tacro (Envarsus®)
Biological: Pharmacocinetik — Nine sampling points of 7 ml each will be taken on the first day at the CIC UIC and the last sampling point will be carried out at 24 hours from the administration the following morning.
Genetic: Genetic — A genetic analysis to determine your characteristics for enzymes in your metabolism as well as transport proteins will be carried out. An additional 7 ml blood tube will be drawn for this purpose during the first period.
Other: Selection visit: — During this visit, it will be asked to sign the following consent and it will be carried out:
  * a clinical examination (questioning and physical examination with measurement of height and weight);
  * a blood test (18 mL);
  * a blood pregnancy test if you are a woman;
  * a cardiac assessment (electrocardiogram).
  These results should be normal.

SUMMARY:
Tacrolimus is a drug administered orally available with different formulations: immediate release (Prograf®), prolonged-release (Advagraf®) and an extended-release one named LCP-Tacro (Envarsus®), formulated using the Melt-Dose process.

Tacrolimus is a lipophilic macrolide drug able to passive transmembrane diffusion. Its bioavailability displays a large interindividual variability, from 9 to 43%. Indeed, tacrolimus is a substrate of P-glycoprotein (P-gp) and cytochrome P450 3A4 (CYP3A4). P-gp is an efflux protein mainly located at the apex of the epithelia of the intestine, lymphocyte, kidney and blood-brain barrier. P-gp therefore limits the intestinal resorption of tacrolimus and also its diffusion into its target compartment (i.e the lymphocyte. The expression of this protein is different throughout the digestive tract with maximum expression at the ileal level. CYP3A4 is a coenzyme that is responsible of more than 90% of the metabolism of tacrolimus, at the digestive and hepatic level. Both P-gp and CYP3A4 play a role in tacrolimus absorption/diffusion process.

A new formulation of tacrolimus, LCP-Tacro, (Envarsus®) was approved in 2014. Its efficacy was compared to Prograf® in two phase III de novo or switch Prograf® trials in kidney transplantation.

With tacrolimus, there is a strong inter-individual pharmacokinetic variability which, to date, has not been fully characterized. Variations in bioavailability may partly explain this high variability. The different formulations are resorbed at distinct gastrointestinal sites which could explain different absorptions between Prograf/Advagraf and LCP-Tacro forms.

These findings raise the question of the role of P-gp in explaining the difference in bioavailability between formulations. The use of a P-gp inhibitor could therefore have a different impact on exposure to different galenic formulations.

Verapamil is an inhibitor of P-gp and CYP 3A4, which is frequently prescribed and recommended by FDA for drug-drug interaction studies aiming at evaluating P-gp substrates, used in healthy volunteers at dosages up to 240 mg/D13-14. Otherwise, verapamil-tacrolimus interaction has been characterized in vitro.

It has also been shown that inhibitory effect of verapamil at a single dose of 120 mg administered one hour prior to the administration of a P-gp substrate exhibited an optimum power of inhibition.

The safety of Advagraf® and Envarsus® administrations have already been subjected to several phase I trials in healthy volunteers reinforcing the knowledge of their safety profile.

The aim of the study is to compare the interaction profile of Advagraf® and Envarsus® when co-administered with verapamil in healthy subjects and to provide guidelines on tacrolimus dosage adjustment in such cases.

ELIGIBILITY:
Inclusion Criteria:

* adults (> 18 years)
* Non smokers (for at least 6 months)
* Biological parameters within normal range (blood count, urea, creatinine, AST, ALT, GGT, bilirubine)
* BMI within 18 and 25
* Vaccinated against Covid 19
* Negative urinary and plasma pregnancy test
* Having effective contraception for the duration of the study and for 10 days after the last administration of the study treatment (for women and men of childbearing potential)
* Informed consent

Exclusion Criteria:

* participation to another study with incompatible procedure regarding the French law on research
* Treatment with a drug drug interaction with tacrolimus
* Cardiac rhythm at rest below 50 bpm
* Cardiac issue detected on electrocardiogram
* Cancer or history of cancer
* Chronic infection or history of chronic infection
* Diabetes or history of diabetes
* Hypertension or history of hypertension
* Pregnancy or lactation
* Deprived of liberty (curatorship, guardianship or incarcerate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve | Between 0 and 24 hours
  Change in area under the curve of tacrolimus blood concentrations between 0 and 24h.

SECONDARY OUTCOMES:
Cmax | Cmax Advagraf: 2-3 hours, Cmax Envarsus: 6-8 hours
  Blood pharmacokinetic parameters: peak concentration (Cmax)
Trough concentration | 24 hours
  Blood pharmacokinetic parameters: trough concentration (Cmin)
Apparent clearance | 0-24 hours
  Blood pharmacokinetic parameters: apparent clearance (Cl/F)
Half-life | 0-24 hours
  Blood pharmacokinetic parameters: half-life (T1/2)).
AUC | 0-24 hours
  Intracellular pharmacokinetic parameters: AUC
Cmax | Cmax Advagraf: 2-3 hours, Cmax Envarsus: 6-8 hours
  Intracellular pharmacokinetic parameters: Cmax
Cmin | 24 hours
  Intracellular pharmacokinetic parameters:Cmin
CI/F | 0-24 hours
  Intracellular pharmacokinetic parameters: Cl/F
T1/2 | 0-24 hours
  Intracellular pharmacokinetic parameters:T1/2
ABCB1 genotypes | Day 0
  ABCB1 genotypes
Others genotypes | Day 0
  Other genotypes of interest coding for metabolism (CYP3A4, CYP3A5…) or drug transport (CNT3…).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France